CLINICAL TRIAL: NCT01387724
Title: Neuropeptide Y and Its Receptors in Neuroblastoma
Brief Title: Biomarkers in Blood and Tissue Samples From Patients With Newly Diagnosed Neuroblastoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ANBL11B1; COG-ANBL11B1 (Other: Children's Oncology Group); NCI-2011-02862 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ANBL11B1 (Other: Children's Oncology Group)
Record Dates: First submitted 2011-07-01; First posted 2011-07-04 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Neuroblastoma
Keywords: disseminated neuroblastoma; localized resectable neuroblastoma; localized unresectable neuroblastoma; regional neuroblastoma; stage 4S neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Polymerase Chain Reaction; Blotting, Western; Enzyme-Linked Immunosorbent Assay; Immunohistochemistry; Chromatography, Liquid; Mass Spectrometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and tissue
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: RNA analysis
Genetic: polymerase chain reaction
Genetic: protein expression analysis
Genetic: proteomic profiling
Genetic: western blotting
Other: enzyme-linked immunosorbent assay
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Other: liquid chromatography
Other: mass spectrometry

SUMMARY:
RATIONALE: Studying samples of blood and tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research trial studies biomarkers in blood and tissue samples from patients with newly diagnosed neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the expression of neuropeptide Y (NPY) and its receptors (Rs) in human neuroblastoma (NB) tissues.
* Determine whether BDNF/TrkB and TrkAIII stimulate expression of NPY and its Rs.
* Determine whether NPY mediates BDNF- and TrkAIII-induced NB proliferation and survival.
* Determine neurotrophins' angiogenic actions.
* Identify factors released from NB cells upon NPY stimulation (proteomics).
* Determine whether NPY upregulates expression of the identified proteins in NB and their Rs in endothelial cells (ECs).
* Test whether inhibition of the identified pathways reduces angiogenic activity of NB-conditioned media.
* Determine the mechanisms of NYP actions and signaling pathways.
* Test whether blocking NPY-Y2/Y5 pathway reduces NB growth and vascularization in vivo.

OUTLINE: Archived tumor tissue and serum samples are analyzed for neuropeptide Y and its receptors (Y1, Y2, and Y5) expression, neuroblastoma prognostic factors (MYCN, TrkA, TrkAIII, TrkB, BDNF, and NGF), and angiogenic markers by real-time PCR, IHC, ELISA, radioimmunoassay (RIA), mitogenic assay, caspase 3/7 activity assay, western blots, liquid chromatography, tandem mass spectrometry, proteomic assays, and other assays. Results are then analyzed and compared with patients' clinical data, including stage of disease, its phenotype, prognostic markers, age and gender, and response to treatment.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Children with newly diagnosed neuroblastoma or ganglioneuroblastoma
* Samples from the Children's Oncology Group (COG) from patients enrolled in clinical trials in institutions in the USA, Canada, and Australia

  * Paraffin-embedded tumor specimens, RNA isolated from tumor tissues, and patient serum must be available

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with newly diagnosed neuroblastoma or ganglioneuroblastoma.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-06; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Association of high expression of NPY and its Y2/Y5 Rs in NBs with poor outcome of the disease, advanced stage, increased vascularization and other unfavorable prognostic factors, such as TrkB expression and MYCN amplification
BDNF/TrkB and TrkAIII up-regulate expression of NPY and its Rs
NPY upregulates expression of the identified proteins in NB and their Rs in endothelial cells (ECs)
Interaction between Y2 and Y5 receptors in NB and ECs sensitize them to NPY and amplify NPY-induced proliferation
Blocking the NPY-Y2/Y5 pathway reduces NB growth and tumor vascularization

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Kitlinska, PhD, Principal Investigator — Lombardi Comprehensive Cancer Center